CLINICAL TRIAL: NCT05124171
Title: Immunogenicity and Reactogenicity Following a 3rd Dose of COVID-19 mRNA Vaccine (Pfizer-BioNtech) and Two Adjuvanted Sub-unit Vaccines (SP/GSK) Administered as a Booster in Adults Who Received 2 Doses of Pfizer-BioNTech mRNA Vaccine as a Primary Vaccination: A Randomized, Single-blinded Multicenter Clinical Trial
Brief Title: Immunogenicity and Reactogenicity Following a Booster Dose of COVID-19 mRNA Vaccine (Pfizer-BioNtech) and Two Adjuvanted Sub-unit Vaccines (SP/GSK) Administered in Adults Who Received 2 Doses of Pfizer-BioNTech mRNA Vaccine as a Primary Vaccination
Acronym: COVIBOOST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: COVIREIVAC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APHP211184; 2021-004550-33 (EudraCT Number)
Record Dates: First submitted 2021-11-08; First posted 2021-11-17 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Vaccine Reaction
Keywords: COVID 19; mRNA vaccines; Immunology; Sub-unit vaccine; Booster
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comirnaty® (Pfizer-BioNTech) (Experimental): Length of use : 1 day
  Interventions: Biological: BNT162b2
- CoV2 preS dTM adjuvanted vaccine (D614), Sanofi/GSK (Experimental): Length of use : 1 day
  Interventions: Biological: CoV2 preS dTM adjuvanted vaccine (D614), Sanofi/GSK
- CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK (Experimental): Length of use : 1 day
  Interventions: Biological: CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK

INTERVENTIONS:
Biological: BNT162b2 — ARM 1 receiving Pfizer-BioNTech vaccine
  * Group 1.A: 18-64 years old
  * Group 1.B: 65 years and older
  Other Names: pfzer/BioNTech, mARN vaccine,
  Arms: Comirnaty® (Pfizer-BioNTech)
Biological: CoV2 preS dTM adjuvanted vaccine (D614), Sanofi/GSK — ARM 2 receiving SP/GSK subunit D614 vaccine
  * Group 2.A: 18-64 years old
  * Group 2.B: 65 years and older
  Arms: CoV2 preS dTM adjuvanted vaccine (D614), Sanofi/GSK
Biological: CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK — ARM 3 receiving SP/GSK subunit B.1.351 vaccine
  * Group 3.A: 18-64 years old
  * Group 3.B: 65 years and older
  Arms: CoV2 preS dTM adjuvanted vaccine (B.1.351), Sanofi/GSK

SUMMARY:
The vaccination campaign in France began in early 2021 and was declared mandatory for all French people in July 2021. The efficacy of COVID-19 vaccines has since been widely demonstrated, as well as their safety, and now 60% of the adult population in France has received a first dose, most of them with Pfizer-BioNTech's mRNA vaccine.

However, despite the increasing coverage, new data highlight the need for a booster dose for the most vulnerable people, including patients with immune deficiency. This makes it likely that a booster dose will also be needed in the general population, especially among healthcare workers, due to the active circulation of new variants since the beginning of summer 2021 and evidence of reduced protection against them.

On the other hand, in addition to evaluating the potential benefit of a booster vaccination, it appears interesting to also evaluate a heterologous vaccination regimen, i.e. a booster with a different vaccine than the one used for the primary vaccination. Some studies have already evaluated a two-dose heterologous regimen and the results have shown stronger protection against SARS-CoV-2. In addition, this alternative could provide a real benefit in terms of accessibility, cost, and acceptability.

The vaccine developed by Sanofi-Pasteur is based on a traditional recombinant protein approach using GSK's AS03 adjuvant. Two formulations of this vaccine are currently under development, the first targeting the S protein of the D614 strain (Wuhan strain), the second targeting the B.1.351 variant. Their value as a booster needs to be evaluated.

The objective of this trial is therefore to evaluate the immunological response and safety induced by a homologous vaccine booster (Pfizer-BioNTech vaccine booster) and a heterologous vaccine booster (one of the two experimental Sanofi/GSK vaccines booster), on the D614 (Wuhan) strain and on the SARS-CoV-2 variants.

DETAILED DESCRIPTION:
The efficacy of COVID 19 vaccines for reducing the risk of severe COVID-19 infection has now been demonstrated in real life. In France, the vaccination campaign started on December 27th, 2020 and was launched rapidly for healthcare professionals and for individuals at risk of severe COVID on January 2021. On August 5th 30th, 2021, approximately 60% of the population (> 12 years) had already received complete vaccination. Out of approximately 74,3 million doses of vaccine administered, 58 million doses are Pfizer BioNTech vaccine (78%).

Data currently available on the persistence of immunity on the one hand and the appearance of viral variants with reduced sensitivity to vaccine immunity on the other, raise the need to administer further additional dose at an interval from the primary vaccination that remains to be defined, possibly different according to age and co-existing diseases.

Currently, the only data published are related to the administration of a third dose (booster) of the same vaccine as the one used for primary vaccination. However, some vaccines developed more recently could be an interesting alternative for booster dose in terms of reactogenicity, availability, cost and acceptance. Moreover heterologous vaccination could be more immunogenic than homologous scheme.

The vaccine developed by Sanofi Pasteur is based on a conventional adjuvanted recombinant protein approach. Two prototype vaccines are under development, one based on the Spike protein of the SARS CoV-2 D614 strain, the other on the B.1.351 strain. Their interest as booster vaccines needs to be investigated.

The objective of this trial is to assess the response induced by a booster dose of either recombinant protein-based subunit vaccine (targeting D614 strain or B.1.351 strain) or by a booster dose of Pfizer-BioNTech mRNA vaccine (targeting Wuhan strain) in individuals previously vaccinated with 2 doses of Pfizer-BioNTech mRNA vaccine. These results will provide important information for booster vaccination recommendations.

Participants enrolled will be healthy adults with no medical history of COVID-19; they will be recruited in 10(15?) centers in mainland France, via the COVIREIVAC network.

The study will be a randomized, single-blinded, multicentre trial with three parallel arms:

ARM 1 receiving Pfizer-BioNTech vaccine

* Group 1.A: 18-64 years old
* Group 1.B: 65 years and older

ARM 2 receiving SP/GSK subunit D614 vaccine

* Group 2.A: 18-64 years old
* Group 2.B: 65 years and older

ARM 3 receiving SP/GSK subunit B.1.351 vaccine

* Group 3.A: 18-64 years old
* Group 3.B: 65 years and older

Participants will undergo 5 visits :

* V1 (D0): inclusion, randomization, pregnancy test, PCR test, blood draw and administration of the booster dose
* V2 (D28): follow-up visit with a review of solicited and unsolicited local and systemic reactions that occurred since the last visit, and blood draw
* V3 (D90): follow-up visit with review of potential adverse events and blood draw
* V4 (D180): follow-up visit with review of potential adverse events and blood draw
* V5 (D365): follow-up visit with review of potential adverse events and blood draw

Blood samples will be used to conduct immunological analyses, and cellular analyses for a sub-category of 26 participants per group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Adult in a healthy condition or with a stable health status if pre-existing medical history. Stable health status is defined as an existing disease that has not required a significant change in treatment of hospitalization for worsening in the 3 months before enrollment, and for which neither a significant change in treatment or hospitalization for worsening is expected in the near future
3. For women of childbearing age: a negative highly sensitive pregnancy urinary test during the inclusion visit AND use of an effective contraceptive method prior to vaccination and until at least 12 weeks after the vaccination
4. Who has received 2 doses of mRNA vaccine (Pfizer-BioNTech) with an interval of 3 to 6 weeks
5. Second dose of mRNA vaccine (Pfizer-BioNTech) administered 6 months +/- 1 month before the booster dose
6. Understands and agrees to comply with the study procedures
7. Written informed consent signed by both the participant and the investigator
8. Subject affiliated to the French Social Security System.

Exclusion Criteria:

1. Acute febrile infection (body temperature ≥ 38.0°C) within the previous 72 hours and/or presenting symptoms suggestive of COVID-19 within the previous 28 days, or having been in contact with an infected individual for the last 10 days before the inclusion visit;
2. Virologically documented history of COVID-19 (PCR or serology);
3. Immunosuppressive therapy such as corticosteroids > 10 mg prednisone equivalent/day (excluding topical preparations and inhalers) within 3 months prior to inclusion or within 6 months for chemotherapies;
4. Treatment with immunoglobulins or other blood derivatives within 3 months prior to inclusion or scheduled administration of immunoglobulins or blood derivatives before the end of the study;
5. Known HIV, HCV or HBV infection;
6. Any medical condition, such as cancer, that might impair the immune response;
7. Use of experimental immunoglobulins, experimental monoclonal antibodies or convalescent plasma is not permitted during the study;
8. Pregnancy or breastfeeding currently ongoing;
9. History of severe adverse events following vaccine administration including anaphylactic reaction and associated symptoms such as rash, breathing problems, angioedema, and abdominal pain, or a history of allergic reaction that could be triggered by a component of the SARS-COV-2 vaccine at the time of the first vaccine injection;
10. Participant who has received BCG (tuberculosis) vaccine within the previous year;
11. Has received a vaccine within 4 weeks prior to the boost injection or is scheduled to receive a registered vaccine 4 weeks after the boost injection
12. Any bleeding disorder considered as a contraindication to an intramuscular injection, previous phlebotomy, or receipt of anticoagulants
13. Participation in other research involving humans (French classification Jarde 1 or Jarde 2) within 4 weeks prior to the inclusion visit, or participation in any other vaccine trial
14. Subject under legal protection (e.g. guardianship, tutorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
rate of neutralizing antibody titers against SARS-CoV-2 D614 and B.1.351 viral strains | 15 days
  Increased rate of at least 10 fold between D0 and D15 after the booster dose in neutralizing antibody titers against SARS-CoV-2 D614 and B.1.351 viral strains, measured by a microneutralisation technique in each group to assess the immunogenicity of a booster dose of an adjuvanted subunit vaccine (SP vaccine) as between D614 or B.1.351 and a mRNA vaccine (Pfizer BioNTech) in adults who were primarily vaccinated with 2 doses of mRNA vaccine (Pfizer BioNTech) with the 2nd dose of vaccine received at least 6 months +/- 1 month prior to the booster dose.

SECONDARY OUTCOMES:
Rate of increase in neutralizing antibody titers against SARS-CoV-2 D614 and B.1.351 viral strains | 28 days
  Rate of increase in neutralizing antibody titers against SARS-CoV-2 D614 and B.1.351 viral strains, measured by a microneutralisation technique between 0 and 28 days after the booster dose in each group
Quantity and intensity of unsolicited local and systemic events up to 7 days | 7 days
  Quantity and intensity of local and systemic events of any grade occurring up to 7 days after boost injection (assessed from the list of solicited adverse events)
Quantity and intensity of unsolicited local and systemic events up to 28 days | 28 days
  Quantity and intensity of local and systemic events of any grade occurring up to 28 days after boost injection (assessed from the list of solicited adverse events)
Anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels | between Month 3 and Day 0
  Anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels, expressed in BAU/ml, according to WHO recommendations D28 after the booster dose mRNA or adjuvanted subunit vaccine
Difference in anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels at 3 months | Between Month 6 and Day 0
  Difference in anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels between M3 and D0
Difference in anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels at 12 months | between Month 12 and Day 0
  Difference in anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels between M12 and D0
Neutralizing antibody titers against D614, alpha, gamma and delta variants at 3 months | 3 months
  Neutralizing antibody titers against D614, alpha, gamma and delta variants at 3 months
Neutralizing antibody titers against D614, alpha, gamma and delta variants at 3 months | 6 months
  Neutralizing antibody titers against D614, alpha, gamma and delta variants at 3 months
Neutralizing antibody titers against D614, alpha, gamma and delta variants at 12 months | 12 months
  Neutralizing antibody titers against D614, alpha, gamma and delta variants at 12 months
ELISpot IFN CD4 and CD8 response at 28 days | 28 days
  ELISpot IFN CD4 and CD8 response at 28 days
ELISpot IFN CD4 and CD8 response at 3 months | 3 months
  ELISpot IFN CD4 and CD8 response at 3 months
ELISpot IFN CD4 and CD8 response at 12 months | 12 months
  ELISpot IFN CD4 and CD8 response at 12 months
Anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels | Day 3
  Anti-Spike (D614) and anti-RBD (D614 and B.1.351) IgG levels, expressed in BAU/ml, according to WHO recommendations D3 after the booster dose mRNA or adjuvanted subunit vaccine (ancillary analysis) to assess the early humoral response by ELISA of a booster dose of mRNA vaccine or subunit adjuvanted vaccine
ELISpot IFN CD4 and CD8 response | 28 days, 3 months and 12 months
  ELISpot IFN CD4 and CD8 response (ancillary analysis); to explore CD4 and CD8 cellular response induced by a booster dose of mRNA vaccine or adjuvanted subunit vaccine (ancillary analysis)
Activated (CD71+) spike Beta specific B cells will also be sorted and cultured in single cells for further analysis of their BCR and their relationship with the early CSA response. | Day 3
  To explore B cells (CD71) functionality
  Ancillary study endpoints:
  Cf. Coviboost ancillary study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- GH Broca-Cochin-Hôtel-Dieu CIC 1417 Cochin-Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No